CLINICAL TRIAL: NCT03056339
Title: Dose Escalation Study Phase I/II of Umbilical Cord Blood-Derived CAR-Engineered NK Cells in Conjunction With Lymphodepleting Chemotherapy in Patients With Relapsed/Refractory B-Lymphoid Malignancies
Brief Title: Umbilical & Cord Blood (CB) Derived CAR-Engineered NK Cells for B Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0641; NCI-2018-01221 (Registry Identifier: NCI CTRP-Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: B-Lymphoid Malignancies; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Non-hodgkin Lymphoma
Keywords: B-Lymphoid Malignancies; Relapsed/Refractory; Acute lymphocytic leukemia; ALL; Chronic lymphocytic leukemia; CLL; Non-Hodgkin lymphoma; NHL; (CAR).CD19-CD28-zeta-2A-iCasp9-IL15-transduced cord blood natural killer cells; CB-NK cells; Fludarabine; Fludarabine phosphate; Fludara; Cyclophosphamide; Cytoxan; Neosar; AP1903; Mesna; Mesnex
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Recurrence | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna; AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide + CAR-NK Cells (Experimental): On Days -5, -4, and -3, participants receive Fludarabine and Cyclophosphamide. Participants also receive Mesna before and after the cyclophosphamide dose.
  On Day 0, participants receive genetically modified NK cells as a cell infusion.
  If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they receive AP1903 by vein and possibly steroids by mouth or by vein.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Biological: iC9/CAR.19/IL15-Transduced CB-NK Cells; Drug: AP1903

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2 by vein on Days -5 to -3.
  Other Names: Fludarabine phosphate; Fludara
Drug: Cyclophosphamide — 300 mg/m2 by vein on Days -5 to -3.
  Other Names: Cytoxan; Neosar
Drug: Mesna — 300 mg/m2 by vein on Days -5 to -3 before and after the cyclophosphamide dose.
  Other Names: Mesnex
Biological: iC9/CAR.19/IL15-Transduced CB-NK Cells — Infusion of iC9/CAR.19/IL15-transduced CB-NK cells on Day 0 by vein.
  Starting dose: 10E5
  Other Names: NK cells
Drug: AP1903 — If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they will receive AP1903 0.4 mg/kg administered as an intravenous infusion.

SUMMARY:
If you are reading and signing this form on behalf of a potential participant, please note: Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this clinical research study is to learn if giving genetically changed immune cells, called CAR-NK cells, after chemotherapy will improve the disease in stem cell transplant patients with relapsed (has returned) and/or refractory (has not responded to treatment) B-cell lymphoma or leukemia. Also, researchers want to find the highest tolerable dose of CAR-NK cells to give to patients with relapsed or refractory B-cell lymphoma or leukemia. The safety of this treatment will also be studied.

This is an investigational study. The making of and infusion of genetically changed NK cells and the drug AP1903 (if you receive it, explained below) are not FDA approved or commercially available for use in this type of disease. They are currently being used for research purposes only. The chemotherapy drugs in this study (fludarabine, cyclophosphamide, and mesna) are commercially available and FDA approved.

Up to 36 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

To determine the safety and relative efficacy of Chimeric antigen receptors (CAR).CD19-CD28-zeta-2A-iCasp9-IL15-transduced cord blood natural killer (CB-NK) cells in patients with relapsed/refractory CD19+ B lymphoid malignancies.

Secondary Objectives:

1. To assess the overall response rate (complete and partial response rates).
2. To quantify persistence of infused allogeneic donor CAR-transduced CB-derived NK cells in the recipient.
3. To conduct comprehensive immune reconstitution studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of CD 19 positive B-lymphoid malignancies (ALL, CLL, NHL) who have received at least 2 lines of standard chemoimmunotherapy or targeted therapy and have persistent disease.
2. Patients with ALL, CLL, NHL with relapsed disease following standard therapy or a stem cell transplant.
3. Patients at least 3 weeks from last cytotoxic chemotherapy at the time of starting lymphodepleting chemotherapy. Patients may continue tyrosine kinase inhibitors or other targeted therapies until at least two weeks prior to administration of lymphodepleting chemotherapy.
4. Karnofsky/Lansky Performance Scale > 70.
5. Adequate organ function: a. Renal: Creatinine clearance (as estimated by Cockcroft Gault) >/= 60 cc/min. b. Hepatic: ALT/AST </= 2.5 x ULN or </= 5 x ULN if documented liver metastases, Total bilirubin </= 1.5 mg/dL, except in subjects with Gilbert's Syndrome in whom total bilirubin must be </= 3.0 mg/dL. c. Cardiac: Cardiac ejection fraction >/= 50%, no evidence of pericardial effusion as determined by an ECHO or MUGA, and no clinically significant ECG findings. d. Pulmonary: No clinically significant pleural effusion, baseline oxygen saturation > 92% on room air.
6. Able to provide written informed consent.
7. 7-80 years of age.
8. All participants who are able to have children must practice effective birth control while on study. Acceptable forms of birth control for female patients include: hormonal birth control, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence, for the length of the study. If the participant is a female and becomes pregnant or suspects pregnancy, she must immediately notify her doctor. If the participant becomes pregnant during this study, she will be taken off this study. Men who are able to have children must use effective birth control while on the study. If the male participant fathers a child or suspects that he has fathered a child while on the study, he must immediately notify his doctor.
9. Signed consent to long-term follow-up protocol PA17-0483.

Exclusion Criteria:

1. Positive beta HCG in female of child-bearing potential defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females.
2. Known positive serology for HIV.
3. Presence of Grade 3 or greater toxicity from the previous treatment.
4. Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management. Note: Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
5. Presence of active neurological disorder(s).
6. Concomitant use of other investigational agents.

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Nastoupil, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Marin D, Li Y, Basar R, Rafei H, Daher M, Dou J, Mohanty V, Dede M, Nieto Y, Uprety N, Acharya S, Liu E, Wilson J, Banerjee P, Macapinlac HA, Ganesh C, Thall PF, Bassett R, Ammari M, Rao S, Cao K, Shanley M, Kaplan M, Hosing C, Kebriaei P, Nastoupil LJ, Flowers CR, Moseley SM, Lin P, Ang S, Popat UR, Qazilbash MH, Champlin RE, Chen K, Shpall EJ, Rezvani K. Safety, efficacy and determinants of response of allogeneic CD19-specific CAR-NK cells in CD19+ B cell tumors: a phase 1/2 trial. Nat Med. 2024 Mar;30(3):772-784. doi: 10.1038/s41591-023-02785-8. Epub 2024 Jan 18. PMID 38238616
- [Derived] Liu E, Marin D, Banerjee P, Macapinlac HA, Thompson P, Basar R, Nassif Kerbauy L, Overman B, Thall P, Kaplan M, Nandivada V, Kaur I, Nunez Cortes A, Cao K, Daher M, Hosing C, Cohen EN, Kebriaei P, Mehta R, Neelapu S, Nieto Y, Wang M, Wierda W, Keating M, Champlin R, Shpall EJ, Rezvani K. Use of CAR-Transduced Natural Killer Cells in CD19-Positive Lymphoid Tumors. N Engl J Med. 2020 Feb 6;382(6):545-553. doi: 10.1056/NEJMoa1910607. PMID 32023374
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 2017 to May 2021. All participants were registered at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Patient accession #3 and #21 are the same patient. The patient was taken off protocol and re-consented for a second infusion. Patient was only evaluated in regards to safety and efficacy as 1 subject.
Groups:
- Group 1: 1x105 NK Cells /kg: On Days -5, -4, and -3, participants receive Fludarabine and Cyclophosphamide. Participants also receive Mesna before and after the cyclophosphamide dose.
  On Day 0, participants receive genetically modified NK cells as a cell infusion.
  If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they receive AP1903 by vein and possibly steroids by mouth or by vein.
  Fludarabine: 30 mg/m2 by vein on Days -5 to -3.
  Cyclophosphamide: 300 mg/m2 by vein on Days -5 to -3.
  Mesna: 300 mg/m2 by vein on Days -5 to -3 before and after the cyclophosphamide dose.
  iC9/CAR.19/IL15-Transduced CB-NK Cells: Infusion of iC9/CAR.19/IL15-transduced CB-NK cells on Day 0 by vein.
  Starting dose: 10E5
  AP1903: If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they will receive AP1903 0.4 mg/kg administered as an intravenous infusion.
- Group 2: 1x106 NK Cells /kg: On Days -5, -4, and -3, participants receive Fludarabine and Cyclophosphamide. Participants also receive Mesna before and after the cyclophosphamide dose.
  On Day 0, participants receive genetically modified NK cells as a cell infusion.
  If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they receive AP1903 by vein and possibly steroids by mouth or by vein.
  Fludarabine: 30 mg/m2 by vein on Days -5 to -3.
  Cyclophosphamide: 300 mg/m2 by vein on Days -5 to -3.
  Mesna: 300 mg/m2 by vein on Days -5 to -3 before and after the cyclophosphamide dose.
  iC9/CAR.19/IL15-Transduced CB-NK Cells: Infusion of iC9/CAR.19/IL15-transduced CB-NK cells on Day 0 by vein.
  Starting dose: 106
  AP1903: If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they will receive AP1903 0.4 mg/kg administered as an intravenous infusion.
- Group 3: 1x107 NK Cells /kg: On Days -5, -4, and -3, participants receive Fludarabine and Cyclophosphamide. Participants also receive Mesna before and after the cyclophosphamide dose.
  On Day 0, participants receive genetically modified NK cells as a cell infusion.
  If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they receive AP1903 by vein and possibly steroids by mouth or by vein.
  Fludarabine: 30 mg/m2 by vein on Days -5 to -3.
  Cyclophosphamide: 300 mg/m2 by vein on Days -5 to -3.
  Mesna: 300 mg/m2 by vein on Days -5 to -3 before and after the cyclophosphamide dose.
  iC9/CAR.19/IL15-Transduced CB-NK Cells: Infusion of iC9/CAR.19/IL15-transduced CB-NK cells on Day 0 by vein.
  Starting dose: 107
  AP1903: If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they will receive AP1903 0.4 mg/kg administered as an intravenous infusion.
- Group 4: 8x108 Flat NK Cell Dose: On Days -5, -4, and -3, participants receive Fludarabine and Cyclophosphamide. Participants also receive Mesna before and after the cyclophosphamide dose.
  On Day 0, participants receive genetically modified NK cells as a cell infusion.
  If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they receive AP1903 by vein and possibly steroids by mouth or by vein.
  Fludarabine: 30 mg/m2 by vein on Days -5 to -3.
  Cyclophosphamide: 300 mg/m2 by vein on Days -5 to -3.
  Mesna: 300 mg/m2 by vein on Days -5 to -3 before and after the cyclophosphamide dose.
  iC9/CAR.19/IL15-Transduced CB-NK Cells: Infusion of iC9/CAR.19/IL15-transduced CB-NK cells on Day 0 by vein.
  Starting dose: 108
  AP1903: If participant has graft-versus-host disease (GvHD) or cytokine release syndrome after the NK cell infusion, they will receive AP1903 0.4 mg/kg administered as an intravenous infusion.
Period: Overall Study
Arm/Group | Group 1: 1x105 NK Cells /kg | Group 2: 1x106 NK Cells /kg | Group 3: 1x107 NK Cells /kg | Group 4: 8x108 Flat NK Cell Dose
Started | 3 | 6 | 23 | 17
Completed | 3 | 4 | 16 | 16
Not Completed | 0 | 2 | 7 | 1
Not completed — Failed Requirements | 0 | 2 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 1x105 NK Cells /kg | Group 2: 1x106 NK Cells /kg | Group 3: 1x107 NK Cells /kg | Group 4: 8x108 Flat NK Cell Dose | Total
Number analyzed (Participants) | 3 | 6 | 23 | 17 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 11 | 9 | 28
  >=65 years | 0 | 1 | 12 | 8 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 8 | 6 | 18
  Male | 2 | 3 | 15 | 11 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 6 | 21 | 16 | 45
  Unknown or Not Reported | 1 | 0 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 23 | 17 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Events That Was Grade 3-4 Toxicities
Description: Toxicity is defined as a grade 3 or 4 within 40 days of NK cell infusion.
Time Frame: 40 days
Measure: Number; unit: events
Arm/Group | Group 1: 1x105 NK Cells /kg | Group 2: 1x106 NK Cells /kg | Group 3: 1x107 NK Cells /kg | Group 4: 8x108 Flat NK Cell Dose
Number analyzed (Participants) | 3 | 6 | 23 | 17
events
  Grade 3 - Toxicities | 4 | 1 | 22 | 1
  Grade 4 - Toxicities | 0 | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate of Participants Analyzed
Description: Participants response was defined as partial or complete response by Efftox assessment below.
  * Acute lymphoblastic leukemia: Complete response will be defined as bone marrow with < 5% blasts, the absence of circulating blasts, and no extramedullary sites of disease (as assessed by means of computed tomography or positron-emission tomography), regardless of cell-count recovery.
  * CLL: Response will be defined based on the NCI-WG/IWCLL 2008 criteria, Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia.
  Lymphomas: Response will be defined based on the Lugano criteria- Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma:
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Group 1: 1x105 NK Cells /kg | Group 2: 1x106 NK Cells /kg | Group 3: 1x107 NK Cells /kg | Group 4: 8x108 Flat NK Cell Dose
Number analyzed (Participants) | 3 | 6 | 23 | 17
participants
  Complete Response | 2 | 3 | 3 | 5
  Partial Response | 0 | 0 | 5 | 3
  Progressive Disease | 1 | 1 | 6 | 2
  Not Evaluable | 0 | 2 | 7 | 2
  Stable Disease | 0 | 0 | 2 | 5

3. Secondary Outcome: Number of Participants Achieved an Objective Response
Description: Number of participants that had Complete and Partial Response.
Time Frame: Up to 100 days after NK cell infusion
Measure: Number; unit: participants
Arm/Group | Group 1: 1x105 NK Cells /kg | Group 2: 1x106 NK Cells /kg | Group 3: 1x107 NK Cells /kg | Group 4: 8x108 Flat NK Cell Dose
Number analyzed (Participants) | 3 | 6 | 23 | 17
participants
  Complete Response | 2 | 3 | 4 | 5
  Partial Response | 0 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of infusion up to 40 days.
Arm/Group | Group 1: 1x105 NK Cells /kg | Group 2: 1x106 NK Cells /kg | Group 3: 1x107 NK Cells /kg | Group 4: 8x108 Flat NK Cell Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/23 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 0/23 | 0/17
Other Adverse Events (participants affected / at risk) | 2/3 | 6/6 | 12/23 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 1x105 NK Cells /kg (N=3) | Group 2: 1x106 NK Cells /kg (N=6) | Group 3: 1x107 NK Cells /kg (N=23) | Group 4: 8x108 Flat NK Cell Dose (N=17)
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 1x105 NK Cells /kg (N=3) | Group 2: 1x106 NK Cells /kg (N=6) | Group 3: 1x107 NK Cells /kg (N=23) | Group 4: 8x108 Flat NK Cell Dose (N=17)
Abdominal Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Anorexia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - (Other) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood and lymphatic system disorders (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - (Other), specify (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Dizziness (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Encephalopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (Cardiac disorders) | 2 (2) | 0 (0) | 10 (10) | 10 (10)
Fever (General disorders) | 1 (1) | 0 (0) | 8 (8) | 1 (1)
Gastrointestinal disorders (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Infections and infestations (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Investigations - (Other) (Investigations) | 2 (2) | 6 (8) | 3 (3) | 1 (1)
Metabolism and nutrition disorders - (Other) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 12 (12) | 7 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT03056339/Prot_SAP_000.pdf